CLINICAL TRIAL: NCT02276560
Title: Phase II Multicenter Trial of Neoadjuvant Cisplatin and Nab-paclitaxel for (N2) Defined Stage IIIA Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Cisplatin and Nab-paclitaxel for (N2) Defined NSCLC
Acronym: LCCC1407
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to lack of funding.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1407
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Stage IIIA Non-Small Cell Lung Cancer
Keywords: main tumor ranging from less than 3cm (T1 up to 7cm (T3)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Albumin-Bound Paclitaxel; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neoadjuvant Cisplatin,nab-paclitaxel (Experimental): Neoadjuvant cisplatin (75 mg/m2) D1 and nab-paclitaxel (125 mg/m2) D1, 8, 15, repeat each 28D cycle x 3 and then surgery per standard of care
  Interventions: Drug: Neoadjuvant Cisplatin, nab-paclitaxel
- Adjuvant Cisplatin,nab-paclitaxel (Experimental): Adjuvant cisplatin (75mg/m2) D1, nab-paclitaxel (125 mg/m2)for D1, 8, 15 repeat each 28D x 2
  Interventions: Drug: Adjuvant Cisplatin,nab-paclitaxel
- Cisplatin+pemetrexed or gemcitabine (Other): Adjuvant cisplatin (75mg/m2) D1, pemetrexed (500mgm2) D1 or; cisplatin (75 mg/m2),Gemcitabine (1000mg/m2) D1, 8 repeat each 21D cycle x 4
  Interventions: Drug: Adjuvant cisplatin+pemetrexed or cisplatin+gemcitabine

INTERVENTIONS:
Drug: Neoadjuvant Cisplatin, nab-paclitaxel — Cisplatin (75mg/m2) D1, nab-paclitaxel 125 mg/m2) D1, 8, 15; repeat each 28 D cycle x 2 then surgery
  Other Names: Platinol; Abraxane
  Arms: Neoadjuvant Cisplatin,nab-paclitaxel
Drug: Adjuvant Cisplatin,nab-paclitaxel — Cisplatin 75mg/m2 D1,nab-paclitaxel 125mg/m2 D1, 8, 15, repeat each 28D cycle x 2
  Other Names: Platinol; Abraxane
  Arms: Adjuvant Cisplatin,nab-paclitaxel
Drug: Adjuvant cisplatin+pemetrexed or cisplatin+gemcitabine — Cisplatin 75mg/m2 D1 + pemetrexed 500mg/m2 D1 or Gemcitabine 1000 mg/m2 D1, 8 (if SqCC) repeat each 21 D Cycle x 4
  Other Names: Platinol; Alimta; Gemzar
  Arms: Cisplatin+pemetrexed or gemcitabine

SUMMARY:
The purpose of this research study is to determine whether giving cisplatin and nab-paclitaxel before surgery will reduce the presence of disease in certain areas of the lung at the time of surgery.

DETAILED DESCRIPTION:
Objectives

To estimate the rate of N2 nodal clearance at time of surgery in patients with NSCLC undergoing treatment with neoadjuvant nab-paclitaxel plus cisplatin and surgery.

Estimate response rate and complete response rate in non-small cell lung cancer (NSCLC) after 3 cycles of neoadjuvant nab-paclitaxel plus cisplatin

Estimate complete pathological response of primary tumor and lymph nodes at the time of surgery in patients with NSCLC undergoing treatment with neoadjuvant nab-paclitaxel plus cisplatin

Estimate disease free survival for all patients who undergo surgery and also stratified by nodal clearance

Patients will be assigned to receive three (3) cycles of cisplatin (mg/m2) and nab-paclitaxel (125 mg/m2). Surgery will then be conducted per standard of care.

Approximately 4-12 weeks after the surgical resection, patients will receive one of three available treatment regimens based on the results of the surgical reports, which include: Two four week cycles of therapy of Cisplatin and Nab-paclitaxel; Four three-week cycles of Cisplatin and Pemetrexed, or four three-week cycles of Cisplatin and Gemcitabine

Thirty (30) days after treatment ends, subjects will be followed for any ongoing serious adverse events, if necessary, and every 3-6 months thereafter for two years.

After the two years of follow-up, subjects will be followed for survival and disease status

Estimate overall survival for entire group and stratified by nodal clearance

To estimate event free survival (EFS)

Estimate time to distant recurrence and time to local recurrence following total study procedures

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age; no upper age limit
* Diagnosis of NSCLC, histologically or cytologically confirmed
* Pathologic mediastinal staging to include endobronchial ultrasound with or without endoscopic ultrasound (EBUS =/- EUS) including evaluation of N3 nodes
* Systemic staging including CT that covers the chest, liver and adrenal glands or a PET/CT; MRI of the brain is required and must be negative for metastatic spread. If a patient is unable to tolerate MRI or has a contraindication to MRI, a head CT scan with and without contrast is acceptable
* International Association for the Study of Lung Cancer (IASLC) version 7, subset of stage IIIA single station (N2) disease; specifically T1a-T3, N2(+) with no invasion of key structures (e.g., chest wall or diaphragm)
* Surgically resectable disease, and patient deemed an appropriate surgical candidate by a thoracic surgeon prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ and bone marrow function as defined by:

Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Hemoglobin ≥ 10g/dL (it is acceptable to reach this through transfusion); Platelets > 100,000 cells/mm3; Creatinine clearance ≥ 60 mg/dL (Cockcroft-Gault equation); Total bilirubin ≤ 1.5 mg/dL; Alkaline phosphatase ≤ 2.5 x upper limit of normal (ULN); Alanine aminotransferase (ALT, SGPT) ≤ 2.5 x ULN; Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN;

* Women of childbearing potential and sexually active men must agree to use effective contraception prior to study entry, for the duration of study participation and for three months after completing treatment. Adequate contraception is defined as any medically recommended method (or combination of methods) per standard of care
* Negative serum or urine Human Chorionic Gonadotropin(b-hCG) pregnancy test within 14 days of D1 of neoadjuvant chemotherapy for women of childbearing potential
* Informed consent obtained and signed

Exclusion Criteria:

* Forced expiratory volume (FEV) ≤ 1.2 L/s
* T3 tumor defined by invasion of key structures (only T3 defined by size > 7cm allowed)
* Any lymph code > 3 cm or multistation N2 lymphadenopathy
* Patient better served by concurrent chemoradiotherapy: The protocol recognizes that institutional standards regarding which patients are best served by operative and nonoperative approaches vary. Therefore, consistent with the American College of Chest Physicians (ACCP) guidelines, the protocol recommends multidisciplinary discussion of each patient and enrollment only of patients felt best serviced by the approach described herein
* ≥ Grade 2 pre-existing peripheral neuropathy (per CTCAEv4)
* Prior history of hypersensitivity to taxane or platinum therapy. If either agent was previously administered, the patient must have tolerated it well and have recovered from any adverse events
* Recurrent disease or second primary lung cancer (only de novo IIIA disease allowed)
* Other active, invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years; localized squamous cell carcinoma of the skin, basal-cell carcinoma of the skin, carcinoma in-situ of the cervix, or other malignancies requiring locally ablative therapy only will not result in exclusion.
* Prior treatment of any kind for this malignancy
* Have received treatment with any drug that has not received regulatory approval for that indication within the 30 days prior to study entry
* Any serious, uncontrolled medical disorder that would impair the ability of the subject to receive protocol driven therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory - Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Rex Cancer Center and Rex of Wakefield, Raleigh, North Carolina
  - Case Western Reserve University - Seidman Cancer Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials - University of North Carolina - Lineberger Comprehensive Cancer Center — http://unclineberger.org/patientcare/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Cisplatin,Nab-paclitaxel | Adjuvant Cisplatin,Nab-paclitaxel | Cisplatin+Pemetrexed or Gemcitabine
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoadjuvant Cisplatin,Nab-paclitaxel | Adjuvant Cisplatin,Nab-paclitaxel | Cisplatin+Pemetrexed or Gemcitabine | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 67 [67 to 67] |  |  | 67 [67 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of N2 Nodal Clearance
Description: N2 disease is defined as involvement of the ipsilateral mediastinal and/or subcarinal lymph nodes; if disease is cleared form these locations, then there is N2 nodal clearance
Time Frame: 3 Months
Population: The only patient registered before funding was withdrawn could not complete treatment due to adverse events.
Arm/Group | Neoadjuvant Cisplatin,Nab-paclitaxel | Adjuvant Cisplatin,Nab-paclitaxel | Cisplatin+Pemetrexed or Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Neoadjuvant Cisplatin,Nab-paclitaxel | Adjuvant Cisplatin,Nab-paclitaxel | Cisplatin+Pemetrexed or Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Cisplatin,Nab-paclitaxel (N=1) | Adjuvant Cisplatin,Nab-paclitaxel (N=0) | Cisplatin+Pemetrexed or Gemcitabine (N=0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Taste Disturbance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes